CLINICAL TRIAL: NCT04972383
Title: A Prospective,Double-Blind Randomized Controlled Trial Comparing Effect of Autologous Platelet-Rich Plasma Versus Hyaluronic Acid Treatment on Progression of Structural Changes in Knee Osteoarthritis
Brief Title: Comparing Effect of Autologous Platelet-Rich Plasma Versus Hyaluronic Acid Treatment on Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20170062
Record Dates: First submitted 2021-07-06; First posted 2021-07-22 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2021-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Plasma group (Experimental): single injection platelet rich plasma
  Interventions: Combination Product: Platelet Rich Plasma
- Hyaluronic Acid group (Experimental): single injection of hyaluronic acid
  Interventions: Combination Product: Hyaluronic Acid

INTERVENTIONS:
Combination Product: Platelet Rich Plasma — In the Platelet Rich Plasma group, 4mL Platelet Rich Plasma was given.
  Arms: Platelet Rich Plasma group
Combination Product: Hyaluronic Acid — In the Hyaluronic group, 3mLHYAJOINT Plus was given.
  Arms: Hyaluronic Acid group

SUMMARY:
To compare the efficacy and structural change of intraarticular single platelet-rich plasma(PRP) versus novel crosslinked Hyaluronic Acid(HA)(HyajointPlus) for the treatment of early stage knee osteoarthritis(OA). This was a prospective, double-blind, RCT with an allocation ratio of 1:1.

DETAILED DESCRIPTION:
In the PRP group, an Aeon Acti-PRP set was used and an approximately 4-mL PRP volume was yielded and was used in a single-dose treatment. In the HA group, HYAJOINT Plus containing 60 mg of purified sodium hyaluronate was used in a single-dose treatment. All PRP and HA injection syringes were covered with opaque envelop, and the intra-articular injection procedure was performed by the same physician without ultrasound or other imaging guidance.

ELIGIBILITY:
Inclusion Criteria:

1. patients older than 50 years
2. a diagnosis of primary knee osteoarthritis
3. Kellgren-Lawrence (K-L) grading scale smaller than 3
4. both male and female.

Exclusion Criteria:

1. patients younger than 50 years of age
2. K-L grade 3 or more
3. history or active presence of clinically significant inflammatory articular or rheumatic disease other than OA
4. generalized OA
5. the detection of rapidly progressive OA before the start of the trial
6. underwent any previous lower extremity surgery
7. excessive mechanical axis deviation (varus > 5°, valgus > 5°)
8. body mass index larger than 30
9. history or presence of malignant disorders
10. systemic disorders such as diabetes mellitus, severe cardiovascular diseases, hematologic diseases, immune-deficiencies, and infections
11. systematic or intra-articular corticosteroid therapy in the previous 3 months
12. prior treatment with HA in the past 6 months
13. anticoagulants or antiaggregants therapy in the preceding 30 days
14. non-steroidal anti-inflammatory medications in the preceding 7 days
15. platelet count less than 150,000/ml of blood
16. hemoglobin values less than 12g/dL of blood.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
The change of Western Ontario and McMaster Universities Index (WOMAC) score from baseline | Baseline and 1-month, 3-month, 6-month after injection
  The minimum value of Western Ontario and McMaster Universities Index (WOMAC) score is zero and the maximum is 96, whether higher scores mean a worse outcome.

SECONDARY OUTCOMES:
The change of Knee Cartilage Grading System from baseline | Baseline and 1-month, 3-month, 6-month after injection
  The Cartilage Grading System classifies the cartilage from grades 0 to 6 according to parameters of sharpness, clarity and thickness change of the cartilage band. Grade 0 refers to normal and healthy cartilage, while grade 6 refers to severely eroded cartilage, whether higher scores mean a worse outcome.
The change of Knee Cartilage strain ratio from baseline | Baseline and 1-month, 3-month, 6-month after injection
  The strain represents the elasticity. We used the overlying soft tissue as reference. Larger strain ratio means the cartilage is softer, while smaller strain ratio means the cartilage is harder.
The change of MRI Osteoarthritis Knee Score (MOAKS) from baseline | Baseline and 6-month after injection
  Fourteen subregions are defined for scoring of articular cartilage and bone marrow lesions in cluding patella, femur and tibia region. Grade 0 refers to normal and healthy cartilage without loss, while grade 3 refers >75% cartilage full thickness loss, whether higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hsuan-Ti Huang, M.D, Study Chair — Kaohsiung Medical University, Orthopedics Department
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: starting 12 months after publication
Access Criteria: Studies involving platelet rich plasma, hyaluronic acid can contact us for additional information.